CLINICAL TRIAL: NCT06140966
Title: Clinical Study to Evaluate the Safety and Efficacy of Daratumumab and Carfilzomib-based Induction/Consolidation/Maintenance Therapy in Transplant-eligible, Ultra High-risk, Newly Diagnosed Multiple Myeloma
Brief Title: Study to Evaluate the Safety and Efficacy of Daratumumab and Carfilzomib-based Induction/Consolidation/Maintenance Therapy in Transplant-eligible, Ultra High-risk, Newly Diagnosed Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Chunyan Sun, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-KRD20230808
Record Dates: First submitted 2023-11-14; First posted 2023-11-21 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma; Primary Plasma Cell Leukemia; Extramedullary Multiple Myeloma
Keywords: Daratumumab; Carfilzomib; Multiple Myeloma; Ultra High-risk; Primary Plasma Cell Leukemia; Extramedullary Multiple Myeloma; Autologous stem cell transplant; Double hit
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; carfilzomib; Lenalidomide; Dexamethasone; Calcium Dobesilate; Cisplatin; Epirubicin; Cyclophosphamide; Etoposide; Melphalan; Bortezomib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Treatment (Experimental): Pretrial induction chemotherapy (if required): bortezomib, cyclophosphamid, dexamethasone (VCD).
  Induction Chemotherapy: Daratumumab, Carfilzomib,Lenalidomide, Dexamethasone, CisPlatin, epirubicin, Cyclophosphamide and Etoposide (Dara-KRd-PACE).
  Autologous Stem Cell Transplant (ASCT) : Melphalan, ASCT.
  Consolidation: Daratumumab, Carfilzomib, Lenalidomide, Dexamethasone (Dara-KRd).
  Maintenance: Daratumumab, Carfilzomib, and Dexamethasone (Dara-Kd).
  Interventions: Drug: Daratumumab; Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Cisplatin; Drug: epirubicin; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Melphalan; Procedure: ASCT; Drug: bortezomib

INTERVENTIONS:
Drug: Daratumumab — Given by vein: days 1 and 8 of each Induction cycle; days 1 and 15 of each Consolidation cycle; and day 1of each Maintenance cycle.
  Other Names: Darzalex
Drug: Carfilzomib — Given by vein: days 1,2,8 and 9 of each Induction cycle; days 1, 2, 8, 9,15, and 16 of each Consolidation cycle; days 1, 2,15, and 16 of each Maintenance cycle.
  Other Names: Kyprolis
Drug: Lenalidomide — Given by mouth: days 1-7 of each Induction cycle; days 1-14 of each Consolidation cycle.
  Other Names: Revlimid
Drug: Dexamethasone — Given by mouth or by vein: days 1, 8, 15, and 22 of each Induction cycle; days 1, 8, 15, and 22 of each Consolidation cycle; and days 1 and 15 of every cycle during Maintenance
  Other Names: Baycadron
Drug: Cisplatin — Given by vein: days 1-4 of each Induction cycle
  Other Names: Platinol
Drug: epirubicin — Given by vein: days 1-4 of each Induction cycle
  Other Names: Pharmorubicin
Drug: Cyclophosphamide — Given by vein: days 1-4 of each Induction cycle
  Other Names: Cytoxan
Drug: Etoposide — Given by vein: days 1-4 of each Induction cycle
  Other Names: Eposin
Drug: Melphalan — Given by vein: day -1 of Transplant
  Other Names: Alkeran
Procedure: ASCT — day 0 of Transplant
  Other Names: autologous stem cell transplantation
Drug: bortezomib — given by subcutaneous injection: days 1, 4, 8, and 11 of pretrial induction chemotherapy
  Other Names: Velcade

SUMMARY:
This study will assess whether the combination of daratumumab and carfilzomib-based Induction/Consolidation/Maintenance Therapy with ASCT improves the outcome of patients with ultra high-risk, newly diagnosed multiple myeloma

DETAILED DESCRIPTION:
Survival outcomes for patients with newly diagnosed multiple myeloma (MM) have improved substantially in the past decades, due to the introduction of novel therapeutic strategies. Unfortunately, patients with ultra-high-risk MM, including "double-hit" MM, extramedullary MM (EMM), and primary plasma cell leukemia (pPCL), have a significantly worse prognosis and benefit less from current therapeutic strategies. This study aims to investigate whether a treatment regimen combining daratumumab and carfilzomib-based Induction/Consolidation/Maintenance Therapy with autologous stem cell transplantation (ASCT) can improve the survival outcomes of newly diagnosed, transplant-eligible, ultra high-risk multiple myeloma patients. In the study, participants will receive induction therapy with 2-4 cycles of Dara-KRd-PACE, followed by ASCT, 4 cycles of Dara-KRd consolidation, and then maintenance with 12 cycles of Dara-Kd.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have newly diagnosed ultra high-risk disease, as defined by one of the following:1)"Double hit"Multiple Myeloma (≥2 adverse markers: t(4;14), t(14;16), t(14;20), 1q21+, del(17p),p53 mutation) ,2)Extramedullary Multiple Myeloma, 3) primary plasma cell leukemia.
2. Patients must be either untreated or have not received systemic MM therapy. Prior bisphosphonates and localized radiation are allowed.
3. Aged 18 years to 70 years.
4. Fit for intensive chemotherapy and autologous stem cell transplant (at clinician's discretion).
5. Eastern Cooperative Oncology Group (ECOG) score ≤2 before induction chemotherapy.

Exclusion Criteria:

1. No evidence of high-risk disease.
2. Primary diagnosis of Waldenstrom's disease/POEMS syndrome/light chain amyloidosis.
3. Received therapy for multiple myeloma.
4. Prior or concurrent invasive malignancies.
5. Eastern Cooperative Oncology Group (ECOG) score >2 before induction chemotherapy.
6. Clinically significant allergies or intolerance to daratumumab,carfilzomib,lenalidomide, dexamethasone, cisPlatin, epirubicin, cyclophosphamide,melphalan, and etoposide.
7. Participants with contraindication to thromboprophylaxis.
8. Any uncontrolled or severe cardiovascular or pulmonary disease.
9. Platelet count < 50,000/μL, absolute neutrophil count <1000/μL, and haemoglobin <60 g/L before induction chemotherapy.
10. Calculated creatinine clearance <30 mL/min, alanine transaminase (ALT) or aspertate aminotransferase (AST) >3 times upper limit of normal (ULN). Bilirubin >2 times ULN, except in participants with congenital bilirubinemia, such as Gilbert syndrome (direct bilirubin >2.0 times ULN).
11. Known to be seropositive for history of HIV or known to have active hepatitis B or hepatitis C.
12. Ejection fraction by echocardiogram (ECHO) ≥ 45%, pulmonary function studies <50% of predicted on mechanical aspects (Forced Expiratory Volume 1 (FEV1), Forced Vital Capacity (FVC) and diffusion capacity (DLCO) < 50% of predicted.
13. Uncontrolled or severe cardiovascular or pulmonary disease, clinically significant cardiac disease, uncontrolled diabetes mellitus, or other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
14. Known/underlying medical conditions that, in the investigator's opinion, would make the administration of the study drug hazardous.
15. Participant is a woman who is pregnant, or breast feeding, or planning to become pregnant while enrolled in this trial or within at least 6 months after the last dose of trial treatment. Or, participant is a man who plans to father a child while taking part in this trial or within at least 6 months after the last dose of trial treatment.
16. Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 4 weeks before treatment protocol registration or is currently enrolled in an interventional investigational study.
17. Major surgery within 2 weeks before treatment protocol registration or has not fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study. Kyphoplasty or vertebroplasty is not considered major surgery.
18. Known or suspected of not being able to comply with the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-10-20 (Estimated); Study Completion 2027-10-20 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival | 24 months
  2-year Progression-free survival of participants as determined by investigator assessment.

SECONDARY OUTCOMES:
progression-free survival | 36 months
  progression-free survival of participants as determined by investigator assessment.
overall survival | 36 months
  overall survival of participants as determined by investigator assessment.
overall response rate | 36 months
  Overall response rate as determined by the 2016 International Myeloma Working Group (IMWG) Response Criteria for Multiple Myeloma and 2013 IMWG Response Criteria for Plasma cell leukemia by Independent Review Committee (IRC) and investigator assessment.
minimal residual disease negativity rate | 36 months
  Minimal Residual Disease (MRD) negativity rate as assessed by next generation sequencing.
complete response rate | 36 months
  complete response rate as determined by the 2016 International Myeloma Working Group (IMWG) Response Criteria for Multiple Myeloma and 2013 IMWG Response Criteria for Plasma cell leukemia by Independent Review Committee (IRC) and investigator assessment.
duration of minimal residual disease negativity | 36 months
  determined by the 2016 International Myeloma Working Group (IMWG) Response Criteria for Multiple Myeloma and 2013 IMWG Response Criteria for Plasma cell leukemia by Independent Review Committee (IRC) and investigator assessment.
duration of response | 36 months
  determined by investigator assessment.
adverse events | collected until 3 months after treatment completion
  graded according to the Common Terminology Criteria for Adverse Events v5

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided